CLINICAL TRIAL: NCT05462522
Title: A Phase Ib, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple-Ascending Doses of RO7303509 in Participants With Systemic Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of RO7303509 in Participants With Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA43360; 2021-004578-68 (EudraCT Number)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAD Stage (Experimental): Participants will be randomized in a ratio of 4:1 to receive RO7303509 or placebo, as subcutaneous (SC) injection, one time per month for 3 months. You have a 20% chance of getting placebo.
  Interventions: Drug: RO7303509; Drug: Placebo
- OSE Stage (Experimental): Every participant in the OSE stage will receive study drug and no participant will receive placebo. Participants will receive RO7303509 as SC injection at the same dose as that administered during the MAD stage, one time per month for up to a year.
  Interventions: Drug: RO7303509

INTERVENTIONS:
Drug: RO7303509 — RO7303509 will be administered as SC injection monthly, as specified in each treatment group.
Drug: Placebo — RO7303509 matching placebo will be administered as SC injection monthly, during the MAD stage.
  Arms: MAD Stage

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of RO7303509 treatment in participants with systemic sclerosis (SSc) during a multiple-ascending-dose (MAD) portion of the trial. In the MAD phase, increasing doses of study drug will be tested sequentially. For each dose tested, the MAD stage will consist of a treatment period of 12 weeks followed by either a safety follow-up period of 13 weeks or continued treatment in an optional open-label safety extension (OSE) stage of 52 weeks to assess the long-term safety. All patients in the OSE stage will receive RO7303509 and no patient will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the MAD Stage:

* Weight of 45-150 kg at screening
* Diagnosis of SSc, as defined by 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria and ≤ 10 years disease duration from first non-Raynaud's symptom
* Agreement to remain abstinent or use an effective contraceptive method among males and females with childbearing potential for 4 months after last dose of study drug

Inclusion Criteria for the OSE Stage:

* No clinically significant change in eligibility status
* Completion of the MAD and ability to roll over into the OSE within 5 days

Exclusion Criteria:

* Active rheumatic autoimmune disease other than SSc requiring treatment with disease-modifying therapy
* Pulmonary disease with forced vital capacity (FVC) ≤ 50% of predicted
* History or clinical manifestations of significant metabolic, hepatic, renal, pulmonary, cardiovascular, hematologic, gastrointestinal, urologic, neurologic, or psychiatric disorders
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 4 months after the final dose of study drug
* Major surgery within 8 weeks prior to screening, or major planned surgery during the study or within 3 months after the final dose
* Positive hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody test at screening
* Any serious medical condition or abnormality in clinical laboratory tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately 17 months
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Up to approximately 17 months
Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Test Results | Up to approximately 17 months
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters | Up to approximately 17 months

SECONDARY OUTCOMES:
MAD Stage: Maximum Serum Concentration (Cmax) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or early termination (ET) visit
MAD Stage: Area Under the Concentration vs Time Curve (AUC) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or ET visit
MAD Stage: Time to Maximum Concentration (Tmax) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or ET visit
MAD Stage: Total Clearance (CL) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or ET visit
MAD Stage: Volume of Distribution (V) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or ET visit
MAD Stage: Half-Life (t1/2) of RO7303509 | Predose on Day 1 and at multiple timepoints up to Day 113 or ET visit
MAD and OSE Stage: Percentage of Participants With Anti-Drug Antibodies (ADAs) Against RO7303509 | MAD Stage: Predose on Day 1 and at multiple timepoints up to Day 113 (Week 16) or ET visit; OSE Stage: Predose and multiple timepoints up to Week 52; (up to approximately 1.3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (3):
  - Stanford University, Palo Alto, California
  - Hospital For Special Surgery, New York, New York
  - Metroplex Clinical Research Centre, Dallas, Texas
- Argentina (2):
  - Hospital de Alta Complejidad en Red ?El Cruce? Dr. Néstor Kirchner ? S.A.M.I.C., Buenos Aires
  - Clinica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán
- UZ Leuven, Leuven, Belgium
- France (6):
  - Centre Hospitalier Universitaire de Grenoble - Albert Michallon, La Tronche
  - Hopital Cochin, Paris
  - CHU de Bordeaux, Pessac
  - CHRU Rennes, Rennes
  - Hopitaux Universitaires, Strasbourg
  - Hopital Purpan, Toulouse
- Israel (2):
  - Rambam Medical Center - PPDS, Haifa
  - Meir Medical Center, Kfar Saba
- Poland (2):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Zespol Poradni Specjalistycznych REUMED, Lublin
- Portugal (2):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
- The Alliance Medical Sciences Campus, San Juan, Puerto Rico
- Serbia (2):
  - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Military Medical Academy, Belgrade
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Quironsalud Infanta Luisa, Seville
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No